CLINICAL TRIAL: NCT05129774
Title: Concurrent Chemoradiotherapy Sequenced Radical Surgery for Para-aortic Lymph Node Metastasis of Left-sided Colon and Rectal Cancer
Brief Title: Chemoradiotherapy Sequenced Radical Surgery for Colorectal Cancer With PALNM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: V123456
Record Dates: First submitted 2021-10-28; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-10

CONDITIONS: Colorectal Neoplasms Malignant; Lymph Node Excision; Chemoradiotherapy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radical surgery with PALND (Experimental)
  Interventions: Procedure: Radical surgery with PALND
- radical surgery without PALND (Active Comparator)
  Interventions: Procedure: Radical surgery without PALND

INTERVENTIONS:
Procedure: Radical surgery with PALND — sufficient resection margins of the tumor, D3 dissection of the regional lymph nodes and para-aortic lymph node dissection from the bifurcation of iliac artery to the left renal vein via laparoscopic approach
  Arms: radical surgery with PALND
Procedure: Radical surgery without PALND — surgery includes sufficient resection margins of the tumor and D3 dissection of the regional lymph nodes without PALND
  Arms: radical surgery without PALND

SUMMARY:
In left-sided colon and rectal cancer, the occurrence of synchronous para-aortic lymph node metastasis is rare, with the incidence of being approximate 1-2%. Currently, there has been no standard treatment strategy for this situation. The present trial is designed to evaluate the safety and efficacy of para-aortic lymph node dissection for left-sided colon and rectal cancer with synchronous para-aortic lymph node metastasis

ELIGIBILITY:
Inclusion Criteria:

* age at enrollment is ≥ 18 and ≤ 75 years
* ECOG PS 0-1
* histologically confirmed left-sided colon and rectal carcinoma
* synchronous para-aortic lymph node metastases confirmed by PET-CT, and located below the level of renal veins and above the bifurcation of iliac artery
* patients potential to receive surgery and achieve no evidence of disease (NED)
* able to tolerate surgery
* providing written informed consent

Exclusion Criteria:

* local invasion or distant metastasis other than para-aoritc lymph nodes
* history of other malignant tumor
* coupled with severe systematic diseases (recent myocardial infarction, cardiomyopathy, or acute pulmonary infection)
* emergency surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
5-year OS | From date of recruitment until the date of death from any cause, assessed up to 5 years
  5-year overall survival

SECONDARY OUTCOMES:
DFS | From date of recruitment until the date of disease recurrece, assessed up to 5 years
  5-year disease-free survival
LFFS | From date of recruitment until the date of para-aortic lymph node recurrence, assessed up to 3 years
  Local failure free survival
Postoperative complications | From date of surgery until the date of 30 days after surgery
  Postoperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided